CLINICAL TRIAL: NCT03286517
Title: Changes in the Responsiveness of the Hypothalamic-pituitary-gonadal (HPG) Axis to Kisspeptin-10 Administration During Pubertal Transition in Boys
Brief Title: Link Between the Sensitivity of Kisspeptin Signalling and Pubertal Onset in Boys.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ghulam Nabi (Other)
Responsible Party: Sponsor-Investigator, Ghulam Nabi, Mr., Quaid-e-Azam University
Organization: Quaid-e-Azam University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: QuaideAzamU
Record Dates: First submitted 2017-09-11; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Reproductive Physiological Phenomena
Keywords: Puberty, Sexuality
MeSH Terms: conditions — Sexuality | interventions — KISS1 protein, human

STUDY DESIGN:
Intervention Model Description: All the groups were injected with exogenous IV kisspeptin according to the body weight.
Masking Description: All the participants were told for injecting the kisspeptin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Tanner Stage I (Experimental): A 1ml blood sample was obtained for 30 minutes pre and 120 minutes post-kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) injection periods at 30 min intervals (-30, 0, 30, 60, 90, 120). The dose was 9.5 µg/BW.
  Interventions: Biological: Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany)
- Tanner Stage II (Experimental): A 1ml blood sample was obtained for 30 minutes pre and 120 minutes post-kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) injection periods at 30 min intervals (-30, 0, 30, 60, 90, 120). The dose was 11.50 µg/BW.
  Interventions: Biological: Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany)
- Tanner Stage III (Experimental): A 1ml blood sample was obtained for 30 minutes pre and 120 minutes post-kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) injection periods at 30 min intervals (-30, 0, 30, 60, 90, 120). The dose was 12.67 µg/BW.
  Interventions: Biological: Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany)
- Tanner Stage IV (Experimental): A 1ml blood sample was obtained for 30 minutes pre and 120 minutes post-kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) injection periods at 30 min intervals (-30, 0, 30, 60, 90, 120). The dose was 15.11 µg/BW.
  Interventions: Biological: Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany)
- Tanner stage V (Experimental): A 1ml blood sample was obtained for 30 minutes pre and 120 minutes post-kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) injection periods at 30 min intervals (-30, 0, 30, 60, 90, 120). The dose was 20.5 µg/BW.
  Interventions: Biological: Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany)
- Adult Group (Experimental): A 1ml blood sample was obtained for 30 minutes pre and 120 minutes post-kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) injection periods at 30 min intervals (-30, 0, 30, 60, 90, 120). The dose was 1 µg/kg.
  Interventions: Biological: Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany)

INTERVENTIONS:
Biological: Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) — A neurohormone

SUMMARY:
The specific objective of this study was to investigate the sensitivity of Kisspeptin receptor 1 (KISS1R) by determining the responsiveness of GnRH neuron to kisspeptin administration across the pubertal stages and adult group through measuring plasma LH (luteinizing hormone) and testosterone concentrations.

DETAILED DESCRIPTION:
No studies in humans are available regarding KISS1R signalling that, whether expression of the KISS1 or KISS1R sensitivity increases during the pubertal transition in boys. Kisspeptin regulates HPG (hypothalamic pituitary gonadal) axis by secreting GnRH that acts on the pituitary gonadotrophs to secrete LH and FSH. But in contrast to pubertal period, juvenile period kisspeptin pulsatility is reduced, that leads to low GnRH pulsatility and low level of plasma LH, FSH and testosterone. The objective of this study was to determine the response of exogenous kisspeptin in various juvenile stages up to puberty and also in the adults by measuring the level of plasma LH and testosterone. This study would help us to determine that whether there is any link between the increased sensitivity of kisspeptin signalling and puberty onset?, Or at what Tanner stage pre pubertal boys enter into puberty.

ELIGIBILITY:
Inclusion Criteria:

* Boys were classified into 5 different Tanner stages (I-V) according to the criteria of Feingold D. In Atlas of physical diagnosis. Pediatric endocrinology. 2nd ed. Philadelphia. WB Saunders; 1992, pp. 16-19. For comparison, adult men were also recruited.

Exclusion Criteria:

* Individuals with chronic illness or disorder, i.e. hepatic and renal complications, epilepsy, pneumonia, asthma, orchitis, hernia, cryptorchidism, mental retardation, etc. were excluded from this study

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — children were classified into five pubertal stages called Tanner stages on the basis of a genital examination by a physician.
Enrollment: 30 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2014-08-08 (Actual); Study Completion 2015-03-05 (Actual)

PRIMARY OUTCOMES:
To investigate the sensitivity of KISS1R by determining the responsiveness of GnRH neuron to kisspeptin administration across the pubertal stages and adult group through measuring plasma luteinizing hormone and testosterone concentrations | A time frame for each individual was 3 hours. Kisspeptin-10 was injected intravenously and the blood samples were collected at 30 minutes intervals for 30 minutes pre and 2 hours post kisspeptin-10 injection through cannula.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shahab, PhD, Study Director — Quaid-i-Azam University
Locations (1):
- Quaid-i-Azam University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual response to kisspeptin administration without disclosing the identity of an individual can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: I have already completed the study and can share the data. It will be available in the form of research paper along with the supplementary materials.
Access Criteria: Will be available on journal website after publication or we can share personally.

REFERENCES:
- [Background] Mead EJ, Maguire JJ, Kuc RE, Davenport AP. Kisspeptins are novel potent vasoconstrictors in humans, with a discrete localization of their receptor, G protein-coupled receptor 54, to atherosclerosis-prone vessels. Endocrinology. 2007 Jan;148(1):140-7. doi: 10.1210/en.2006-0818. Epub 2006 Oct 5. PMID 17023533
- [Result] Jayasena CN, Nijher GM, Comninos AN, Abbara A, Januszewki A, Vaal ML, Sriskandarajah L, Murphy KG, Farzad Z, Ghatei MA, Bloom SR, Dhillo WS. The effects of kisspeptin-10 on reproductive hormone release show sexual dimorphism in humans. J Clin Endocrinol Metab. 2011 Dec;96(12):E1963-72. doi: 10.1210/jc.2011-1408. Epub 2011 Oct 5. PMID 21976724
- [Result] Jayasena CN, Nijher GM, Chaudhri OB, Murphy KG, Ranger A, Lim A, Patel D, Mehta A, Todd C, Ramachandran R, Salem V, Stamp GW, Donaldson M, Ghatei MA, Bloom SR, Dhillo WS. Subcutaneous injection of kisspeptin-54 acutely stimulates gonadotropin secretion in women with hypothalamic amenorrhea, but chronic administration causes tachyphylaxis. J Clin Endocrinol Metab. 2009 Nov;94(11):4315-23. doi: 10.1210/jc.2009-0406. Epub 2009 Oct 9. PMID 19820030
- [Derived] Nabi G, Ullah H, Khan S, Wahab F, Duan P, Ullah R, Yao L, Shahab M. Changes in the Responsiveness of the Hypothalamic-Pituitary-Gonadal Axis to Kisspeptin-10 Administration during Pubertal Transition in Boys. Int J Endocrinol. 2018 Jun 26;2018:1475967. doi: 10.1155/2018/1475967. eCollection 2018. PMID 30046307
- Available data/document: Any information required can be provided — http://www.qau.edu.pk/profile.php?id=802001 — Prof. Muhammad Shahab will provide the information upon request.